CLINICAL TRIAL: NCT00891189
Title: Circadian Rhythms and Nocturnal Asthma
Brief Title: Determine the Relationship Between Circadian Rhythms and Nocturnal Asthma
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Phyllis Zee, Professor, Northwestern University
Other Study IDs: 637; K23HL091508 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Circadian Rhythm
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 Control: Healthy participants without asthma
- 2 Non-nocturnal asthma: Participants with non-nocturnal asthma
- 3 Nocturnal asthma: Participants with nocturnal asthma

SUMMARY:
Asthma is a disease that affects the lungs. Symptoms include repeated episodes of wheezing, breathlessness, chest tightness, and nighttime or early morning coughing. Some people with asthma experience worse symptoms at night, which is known as nocturnal asthma (NA). The reason for the decline in lung function at night in some asthmatics is not well understood, but it may be linked to the human biological clock, which controls daily activity and sleep rhythms. To determine whether differences in biological clocks relate to worsening nocturnal lung function, this study will evaluate the circadian rhythms of people with NA, people with non-nocturnal asthma, and healthy people.

DETAILED DESCRIPTION:
Nocturnal worsening of asthma, frequently called NA, is a common problem among some people with asthma and one that leads to increased morbidity and mortality. It is still unknown why lung function worsens at night in some asthmatics and not others. There is a possible relationship between NA, biological clocks, and circadian rhythms, but more research is needed to understand this relationship. Although the diurnal nature of NA has been shown repeatedly in studies, circadian rhythms have not yet been implicated as a related factor. This study will examine the pathophysiology of NA as it relates to circadian biology and will specifically explore physiological and molecular aspects.

This study will include people with asthma, people with NA, and healthy people. Potential participants will attend a screening visit to assess general health and severity of asthma, if present. They will also complete 2 weeks of diary recordings of their daily symptoms and airway function.

Eligible participants will then attend two study visits. The first study visit will last 1 hour and may include a methacholine challenge and bronchodilator testing, both of which will measure lung function. For 2 weeks before the second study visit, participants will keep records of their sleep patterns. The second study visit will be a hospital stay that will last for 2.5 days. While in the hospital, participants will undergo periodic blood draws and lung function testing. During waking hours, participants will remain quietly awake. During the first night, participants will be monitored while they sleep. During the second night, participants will stay awake for 28 hours, which will continue into the third day. Then, on the third day, participants will sleep for 8 hours while again being monitored. Upon waking, participants will be given a regular meal and discharged.

ELIGIBILITY:
Inclusion Criteria for People with Asthma:

* A physician diagnosis of asthma, consistent clinical history, and either 1) airway hyperresponsiveness indicated by a 20% or greater decrease in forced expiratory volume at one second (FEV1) in response to inhalation of methacholine at 8 mg/mL or less, or 2) bronchodilator-responsive expiratory airflow limitation (if FEV1 less than 70% of predicted value or less than 1.5 L, improving at least 200 mL and 12% in response to 180 μg of albuterol aerosol). Patients with NA should meet the above criteria and demonstrate an overnight decrease in peak flow of 20% or greater on at least four of seven nights at home.

Inclusion Criteria for all Participants:

* Able to follow directions

Exclusion Criteria for Participants with Asthma:

* Use of oral steroids within 2 weeks of study entry
* Use of cromolyn, leukotriene antagonist, or theophylline within 1 week of study entry
* History of cognitive or other neurological disorder
* Active symptoms of Diagnostic and Statistical Manual IV (DSM-IV) criteria for any major psychiatric disorder, alcohol abuse, or substance abuse
* History of, or concurrent, unstable or serious medical illness
* Shift work
* History or evidence of chronic obstructive pulmonary disease (COPD)
* Tobacco smoking within the last month, or history of smoking greater than 5 pack-years
* Pregnancy or the desire to become pregnant during the study period
* Hematocrit less than 30
* Worsening or unstable asthma that requires use of a bronchodilator for more than four times a day

Exclusion Criteria for all Participants:

* History of obstructive sleep apnea or a body mass index more than 36, or other sleep disorder as assessed by questioning or polysomnography (PSG)
* History of cognitive or other neurological disorder
* Currently meets DSM-IV criteria for any major psychiatric disorder, alcohol abuse, or substance abuse (as assessed by an interview)
* Concurrent unstable or serious medical illness (other than asthma)
* Current use of psychoactive medications, including antidepressants, anxiolytics, neuroleptics, anticonvulsants, hypnotics, and stimulant medications
* Shift work
* A daily caffeine intake greater than 4 cups per day
* Smoking
* Pregnancy or the desire to become pregnant during the study period
* Atrial fibrillation or paced heart rhythm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy and asthmatic participants
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Spirometry | Measured during the 28-hour constant routine testing

SECONDARY OUTCOMES:
Cortisol, melatonin, exhaled nitric oxide, inflammatory cytokine levels, clock gene expression, and heart rate variability | Measured during the 28-hour constant routine testing

CONTACTS AND LOCATIONS:
Overall Officials: Brandon S. Lu, MD, MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Sutherland ER. Nocturnal asthma. J Allergy Clin Immunol. 2005 Dec;116(6):1179-86; quiz 1187. doi: 10.1016/j.jaci.2005.09.028. Epub 2005 Nov 8. PMID 16337443